CLINICAL TRIAL: NCT01398722
Title: Study of the Relationship Between Intensive Insulin Therapy and Clinical Prognosis in Infants Undergoing Cardiac Surgery
Brief Title: Effect of Intensive Insulin Therapy on Clinical Prognosis of Infants Undergoing Cardiac Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Chunhu Gu, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Guch-012
Record Dates: First submitted 2011-07-11; First posted 2011-07-20 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Cardiac Surgery
Keywords: cardiac surgery; prognosis; intensive insulin therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive insulin therapy (Active Comparator): Intensive insulin therapy(Blood glucose target: 110-150 mg/dL)
  Interventions: Other: Intensive insulin therapy
- Conventional insulin therapy (Active Comparator): Conventional insulin therapy(Blood glucose target: 150-180 mg/dl)
  Interventions: Other: Conventional insulin therapy

INTERVENTIONS:
Other: Intensive insulin therapy — Titration of the IV insulin rate for glucose goal 110-150 mg/dL
  Arms: Intensive insulin therapy
Other: Conventional insulin therapy — Titration of the IV insulin rate for glucose goal 150-180 mg/dl
  Arms: Conventional insulin therapy

SUMMARY:
The investigators sought to determine whether intensive insulin therapy can improve prognosis of infants undergoing cardiac surgery.

DETAILED DESCRIPTION:
Previous studies showed that tight blood glucose control with insulin during intensive care reduced morbidity and mortality of surgical and medical intensive care patients. Blood sugar control with intravenous insulin may improve prognosis of patients undergoing cardiac surgery. It is not clear what the best insulin regimen is or what is the best blood sugar target in these patients. So far, most of researches have focused on adult patients but little on infants. The current prospective, randomized, controlled study will assess the impact of intensive insulin therapy on the outcome of infants undergoing cardiac surgery. On admission, patients will be randomly assigned to either strict normalization of blood glucose ( 110-150 mg/dl) with intensive insulin therapy or the conventional approach, in which blood glucose levels are maintained between 150 and 180 mg/dl.

ELIGIBILITY:
Inclusion Criteria:

* Infants underwent cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* Therapy restricted upon admission
* Preoperative liver or kidney disease or dysfunction
* Preoperative coagulation disorder
* Palliative operation or a second operation
* Type 1 diabetes
* Type 2 diabetes

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 800 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | one year

SECONDARY OUTCOMES:
Biochemical markers of myocardial injury(troponin and creatine kinase MB) | average 1 month during the hospitalization
Acute renal failure | average 1 month during the hospitalization
Respiratory failure | average 1 month during the hospitalization
ICU and hospital length of stay, and ICU readmissions | average 1 month during the hospitalization
Stroke and reversible ischemic neurologic deficit | average 1 month during the hospitalization
Cardiac Index | average 1 month during the hospitalization
Inotropic Scores | average 1 month during the hospitalization
Perioperative complications | average 1 month during the hospitalization
  Perioperative complications including sternal wound infection (deep and superficial), bacteremia, pneumonia, and major cardiovascular events (acute myocardial infarction, congestive heart failure, and cardiac arrhythmias

CONTACTS AND LOCATIONS:
Overall Officials: Dinhhua Yi, MD, Study Chair — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China